CLINICAL TRIAL: NCT04435041
Title: Remote-by-Default Care in the COVID-19 Pandemic: Addressing the Micro-, Meso-, and Macro-level Challenges of a Radical New Service Model
Brief Title: Remote-by-Default Care in the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Plymouth (Other); Nuffield Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 283196
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Remote assessment tools: Qualitative methods: semi-structured interviews for approx 40 front line clinical practitioners
- RECAP early warning score: Development of disease specific early warning score, building on earlier work through literature review and NEWS2 score
- Implementation/Scale up case studies: Study of implementation and scale up of remote-by-default at four different UK sites
- Infrastructure strengthening: Theory and data driven change effort involving policymakers, regulators, professional bodies, industry, patients and citizens with a view to overcoming interacting issues impacting success of digital projects.

SUMMARY:
18 month study, funded by ESRC COVID-19 research fund. The aim is to explore and support the rapid shift from face-to-face to remote (telephone and video) conversations in primary care. There are three components: a study of clinical interactions and decision making (micro); four locality-based organisational case studies of new models of care (meso); abd a a study of how digital innovation can support NHS infrastructure and vice versa (macro).

DETAILED DESCRIPTION:
18 month study, funded by ESRC COVID-19 research fund. The aim is to explore and support the rapid shift from face-to-face to remote (telephone and video) conversations in primary care. There are three components: a study of clinical interactions and decision making (micro); four locality-based organisational case studies of new models of care (meso); abd a a study of how digital innovation can support NHS infrastructure and vice versa (macro). The methods are mainly qualitative (interviews, virtual ethnography, analysis of documents, micro-analysis of conversations) and are designed to inform action research.

Key deliverables:

At least two evidence-based assessment tools: qualitative (questions for remote assessment of breathlessness) and quantitative (a COVID-19-specific early warning score)

Transferable lessons about how to achieve rapid spread and scale-up, spread in real time through our extensive intersectoral networks

Strengthened infrastructure for supporting digital innovation in the NHS

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for interviews

Willing and able to give informed consent for participation

Aged 18 years or above

Staff involved in delivering remote-by-default services in the frontline or 'back offices'

Patients/carers who have crossed paths with primary care services during the Covid pandemic.

Pharmacy case studies:

Staff involved in delivering remote pharmacist consultation services in the frontline or 'back offices'

Patients/carers who have crossed paths with community pharmacy primary care services during the COVID-19 pandemic.

Inclusion criteria for video and telephone consultations

Patients who have remote primary care consultation regarding symptoms associated with COVID-19 and their clinicians (based in Oxford/Thames Valley) who have agreed to participate in the study

Inclusion criteria for focus groups

Patients that have experienced self-reported 'long Covid' symptoms (for patient only focus groups)

Clinicians that have experienced self-reported 'long Covid' symptoms (for clinician only focus groups)

Exclusion Criteria:

Patients or clinicians who are too ill to be interviewed

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mixed methods study
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Remote COVID-19 Assessment in Primary Care (RECAP) Early warning score | 18 months
  A set of questions and a predictive tool built into electronic records, designed to distinguish people with suspected covid-19 who need to go to hospital from those who can safely be monitored at home. The final Remote COVID-19 Assessment in Primary Care (RECAP) Early warning score score divides people into 'green' (stay at home, self-monitor), amber (professional monitoring e.g., via virtual wards with home oximetry), or red (assess in person promptly).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Fiorentino F, Prociuk D, Espinosa Gonzalez AB, Neves AL, Husain L, Ramtale SC, Mi E, Mi E, Macartney J, Anand SN, Sherlock J, Saravanakumar K, Mayer E, de Lusignan S, Greenhalgh T, Delaney BC. An Early Warning Risk Prediction Tool (RECAP-V1) for Patients Diagnosed With COVID-19: Protocol for a Statistical Analysis Plan. JMIR Res Protoc. 2021 Oct 5;10(10):e30083. doi: 10.2196/30083. PMID 34468322
- [Derived] Ladds E, Rushforth A, Wieringa S, Taylor S, Rayner C, Husain L, Greenhalgh T. Persistent symptoms after Covid-19: qualitative study of 114 "long Covid" patients and draft quality principles for services. BMC Health Serv Res. 2020 Dec 20;20(1):1144. doi: 10.1186/s12913-020-06001-y. PMID 33342437
- [Derived] Greenhalgh T, Thompson P, Weiringa S, Neves AL, Husain L, Dunlop M, Rushforth A, Nunan D, de Lusignan S, Delaney B. What items should be included in an early warning score for remote assessment of suspected COVID-19? qualitative and Delphi study. BMJ Open. 2020 Nov 12;10(11):e042626. doi: 10.1136/bmjopen-2020-042626. PMID 33184088

DOCUMENTS (1):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT04435041/Prot_000.pdf